CLINICAL TRIAL: NCT03634891
Title: An Audit Study on Management of Neonates With Neonatal Sepsis Admitted to Asyut University Children Hospital
Acronym: ASMNWNSATAUC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: heba mostafa taher mostafa (Other)
Responsible Party: Sponsor-Investigator, heba mostafa taher mostafa, assiut, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AssiutHM
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Neonates Have Risk Factors or Manifestations of Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study aims to evaluate management of neonates with neonatal sepsis admitted to the Neonatology Unit, Assiut University Children Hospital according to the guidelines of the American Academy of Pediatrics, 2018,[25] searching for defects, obstacles, or needs to improve the management of such cases.

We consider that this critical appraisal of our own performance, is a crucial step before any further corrections or developments of that performance could take place.

DETAILED DESCRIPTION:
Definition:

Neonatal sepsis is a systemic response to infection documented by positive blood culture in the first month of life. [1]

Classification:

It may be categorized as early-onset or late-onset.

Early-onset sepsis is associated with acquisition of microorganisms from the mother. Transplacental infection or an ascending infection from the cervix may be caused by organisms that colonize the mother's genitourinary (GU) tract; the neonate acquires the microorganisms as it passes through the colonized birth canal at delivery. Of newborns with early-onset sepsis, 85% present within 24 hours, 5% present at 24-48 hours, and a smaller percentage present within 48-72 hours. Onset is most rapid in premature neonates. [2]

Late-onset sepsis occurs after 3 days of life and is acquired from the caregiving environment.[3] Pathophysiology:[10] Neonates are particularly vulnerable to infection as a result of lower non-specific immunity (inflammation) and specific (humeral), such as low phagocytosis, chemotaxis response delay, minimal or absence of immunoglobulin A and immunoglobulin M (IgA and IgM), and low levels of complement.

Sepsis in the neonatal period can be obtained before birth through the placenta from the maternal blood stream or during labor for ingestion or aspiration of infected amniotic fluid.

Sepsis early (less than 3 days) obtained in the perinatal period, infection can occur from direct contact with the organism from the gastrointestinal or genitourinary tract maternal. The most frequent infecting organism is group B streptococcus (GBS) and Escherichia coli, which is present in the vagina. GBS emerged as a highly virulent microorganisms in the neonate, with a high mortality rate (50%) in infants exposed to Haemophilus influenzae and Staphylococcus negative coagulation are also often seen in early-onset sepsis in infants with very low birth weight.

Advanced Sepsis (1 to 3 weeks after birth) primarily nosocomial, and organisms that attack is usually staphylococci, Klebsiella, enterococcus and pseudomonas. Coagulation negative staphylococci, commonly found as the cause of septicemia in infants of low birth weight and very low birth weight. Bacterial invasion can occur through such Gated umbilical stump, skin, mucous membranes of eyes, nose, pharynx, and ear, and internal systems such as the respiratory system, nervous, urinary, and gastrointestinal.

Postnatal infection, derived from cross-contamination with other babies, personnel, or objects in the environment. Bacteria commonly found in water sources, a humidifier, sink pipes, suction machines, most equipment respiration, and arterial and venous catheters inserted used for infusion, blood sampling, monitoring of vital signs.

The process begins with the invasion of the pathophysiology of bacterial sepsis and systemic contamination. The release of endotoxin by bacteria cause changes in the function of the myocardium, changes in uptake and utilization of oxygen inhibition of mitochondrial function, and progressive metabolic chaos. In sepsis sudden and severe, complemen cascade caused much death and damage cells. The result is a decrease in tissue perfusion, metabolic acidosis, and shock, disseminated intravascular coagulation resulting (DIC) and death.[11]

Patients with immune disorders have an increased risk for serious nosocomial sepsis. Cardiopulmonary manifestations of gram-negative sepsis can be replicated by injection of endotoxin or Tumor Necrosis Factor (TNF). Barriers to employment TNF by anti-TNF monoclonal antibody greatly weakens manifestation of septic shock. When the bacterialcell wall components are released in the bloodstream, cytokine-activated, and can further lead to more physiological mess. Either alone or in combination, bacterial products and pro-inflammatory cytokines trigger a physiological response to stop the invaders (invader) microbes. TNF and other inflammatory mediators increase vascular permeability and vascular tone imbalance, and the imbalance between perfusion and increased metabolic needs of the network.[12]

Shock is defined as a systolic pressure below the 5th percentile for age or defined with cold extremities. Capillary refilling the late (more than 2 seconds) is seen as a reliable indicator of a decrease in peripheral perfusion. Peripheral vascular pressure in septic shock (heat) but be very up on a further shock (cold). In septic shock tissue oxygen consumption exceeds oxygen supply. This imbalance is caused by peripheral vasodilatation in the beginning, during further vasoconstriction, myocardial depression, hypotension, ventilator insufficiency, and anemia.[13]

Septicemia shows the emergence of a systemic infection of the blood caused by the rapid multiplication of microorganisms or toxic substances, which can cause huge psychological change. These substances can be pathogenic bacteria, fungi, viruses, and rickets. The most common cause of septicemia is a gram-negative organisms. If the protection of the body is not effective in controlling the invasion of microorganisms, septic shock may occur, which is characterized by hemodynamic changes, imbalance of cellular functions, and multiple system failures.

ELIGIBILITY:
Inclusion Criteria:

* 1. All neonates have risk factors of sepsis. 2. All neonates have manifestations of sepsis.

Exclusion Criteria:

* 1. Infants aged more than 28 days.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Medical records of neonates with neonatal sepsis admitted to the Neonatology Unit, Assiut University Children's Hospital during the period from the 1st of January, 2018 to the 31st of December, 2018. These records will be collected and reviewed to choose the cases which fulfilled the inclusion criteria of the study.
  A structured data collection form will be designed to gather the clinical, laboratorial, imaging and therapeutic data from the included records. This form will be designed according to the published guidelines for neonatal sepsis by the American Academy of Pediatrics, 2018. [25] The data will be tabulated using Epi Info, version 16.0, and the results will be examined by Chi-square statistics. The magnitude of significant associations will be presented as p-value, Odds Ratios (OR), and 95% confidence interval for the OR. A p-value of less than 0.05 will be considered statistically significant.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Guidelines of management of Neonatal sepsis According to American Academy of Pediatrics | one year
  outcome of neonates with neonatal sepsis managed according to these guidlines

CONTACTS AND LOCATIONS:
Overall Officials: heba M taher, M. B. B. CH, Principal Investigator — Asyut University Children Hospital
Locations (1):
- Asyut University Children Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No